CLINICAL TRIAL: NCT05409092
Title: Influence of Astaxanthin Supplementation on Exercise-Induced Inflammation and Skin Health
Brief Title: Astaxanthin, Exercise Inflammation, Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: LycoRed Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 22-0100
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Inflammatory Response; Metabolic Disturbance; Immune Suppression
Keywords: astaxanthin; exercise; immune function; proteomics; cytokines; muscle damage
MeSH Terms: conditions — Motor Activity | interventions — astaxanthine

STUDY DESIGN:
Intervention Model Description: Randomized treatment, double blinded procedures, crossover
Who Masked: Participant, Investigator
Masking Description: Investigators and study participants will be blind to treatment allocation, with the astaxanthin and placebo supplements contained in identical looking capsules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astaxanthin (Experimental): The astaxanthin capsules will contain 8 mg of astaxanthin from freshwater algae in starch beadlets. Ingested daily for 4 weeks.
  Interventions: Dietary Supplement: Astaxanthin
- Placebo (Placebo Comparator): The placebo capsules will contain just the starch beadlets with natural red coloring from the pitaya fruit. Ingested daily for 4 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Astaxanthin — 8 mg/day in one capsule for 4 weeks
  Arms: Astaxanthin
Dietary Supplement: Placebo — 8 mg/day in one capsule for 4 weeks
  Arms: Placebo

SUMMARY:
Vigorous exercise can stress the body. Consuming special types of diet supplements may help the body recover better from exercise. This includes a bright red supplement called astaxanthin that is found in certain algae and causes the pink-red color in salmon. Astaxanthin is an antioxidant and may protect cells from damage and improve the way the immune system functions. The main purpose of this study is to determine if 4 weeks of consuming astaxanthin improves recovery from 2.25 hours of intensive running on a treadmill. This study will also measure whether or not astaxanthin supplementation improves skin health

DETAILED DESCRIPTION:
RESEARCH PROCEDURES The research procedures will be conducted at the Human Performance Laboratory (Room 1201, Plants for Human Health Institute Building, 600 Laureate Way), operated by Appalachian State University at the North Carolina Research Campus (NCRC) in Kannapolis, NC. Subjects will come to the Human Performance Lab (HPL) for orientation/baseline testing with pre-supplementation blood sample collections, two 2.25 h running sessions, and additional lab visits to provide 1-day 7:00 am recovery blood samples) (thus 6 total performance lab visits). Skin health measurements will occur the morning before and during Performance Lab Visits #1, 2, 4, 5 (thus 8 total visits, with four of them occurring with HPL visits and four of them occurring separately). The total amount of time subjects will be asked to volunteer for this study is about 16 hours at the North Carolina Research Campus (over a 10-week period).

Orientation/Baseline Testing (Performance Lab Visit #1) Four weeks prior to the first 2.25 h running session, subjects will report to the Human Performance Laboratory at approximately 7:00-8:30 am. Skin health measurements will be conducted the day before (following review of the consent form, with signing) and the day of baseline testing. Following the second skin health measurement, demographic and training histories will be acquired with questionnaires. A symptom inventory will be conducted using a 4-week retrospective questionnaire. Delayed onset of muscle soreness (DOMS) and the Profile of Mood States (POMS) will be assessed with standardized questionnaires. A blood sample will be collected in an overnight fasted state to coincide with the same time of the day for the post-supplementation blood draw. Body composition will be measured with the seca BIA and Bod Pod body composition analyzer (Life Measurement, Concord, CA). Study participants will be tested for maximal aerobic capacity (VO2max) during a graded, treadmill test with the Cosmed CPET metabolic device (Cosmed, Rome, Italy). Supplements for the 4-week supplementation period will be supplied in food supplement trays to facilitate compliance to the supplementation protocol. 3-day food records and the food list will be supplied with thorough instructions (for the 3-day period prior to the 2.25 hour treadmill running sessions).

4-Week Supplementation Periods Study participants will be randomized to astaxanthin and placebo groups, with supplements ingested daily (with the first meal) for 4-weeks prior to participation in the first 2.25 h running session. To assess potential adverse effects, a symptom inventory will be conducted using a 4-week retrospective questionnaire before and after the 4-week supplementation period. After a 2-week washout period, participants will repeat all procedures using the counterbalanced supplement. The astaxanthin and placebo supplements will look identical and be supplied by the sponsor. The astaxanthin capsule will contain 8 mg of astaxanthin from freshwater algae in starch beadlets, and the placebo capsules will contain just the starch beadlets with natural red coloring from the pitaya fruit. Four ounces of sockeye salmon contains about 4.5 milligrams of astaxanthin, with much higher levels in arctic shrimp and krill. Natural astaxanthin is sold around the world as a natural antioxidant supplement with a recommended dosage of 4 mg to 12 mg a day. LycoRed sources astaxanthin from Haematococcus pluvialis, a freshwater algae species of Chlorophyta from the family Haematococcaceae. This species is well known for its high content of the strong antioxidant astaxanthin, which is important in aquaculture, and cosmetics.

2.25 h Running Session (Performance Lab Visit #2, Skin Health Tests #3, #4) During the 3-day period prior to the 2.25 h running session, subjects will taper exercise training and ingest a moderate-carbohydrate diet using a food list restricting high fat foods, visible fats, and polyphenols. Subjects will record all food and beverage intake during the 3-day period, with macro- and micro-nutrient intake assessed using the Food Processor dietary analysis software system (ESHA Research, Salem, OR).

Skin health measurements will be conducted the day before and the day of the running session (#3, #4) (overnight fasted state). Study participants will report to the Human Performance Lab in an overnight fasted state, take the skin health tests, provide a blood sample, ingest astaxanthin or the placebo supplement with water, then run 2.25 h at high intensity (70% VO2max) while ingesting water alone (3 ml/kg every 15 minutes). Blood samples will be collected at 0 h, 1.5 h, 3 h, and 21 h post-exercise.

2-WEEKS WASHOUT, CROSSOVER, REPEAT Subjects will engage in a 2-week washout period without supplements, crossover, and then repeat all procedures (Skin tests #4 through #8; Performance Lab visits #4,5,6). NOTE: Subjects randomized during the first trial to astaxanthin will have 6 weeks of washout when counting the 4-week placebo period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 18-57 years.
* Non-smoker.
* Capable of running 2.25 h on laboratory treadmills at 70% VO2max (close to marathon race pace).
* Agree to train normally, maintain weight, and avoid the regular use of large-dose vitamin and mineral supplements, herbs, and medications that influence inflammation and immune function (especially Advil, Motrin, aspirin, and similar anti-inflammatory drugs) for the duration of the 10-week study. (Review supplement and medication use with the Research Manager during orientation).
* Agree to taper exercise training prior to each of the two lab running sessions (as if preparing for a race).
* Willing to avoid astaxanthin supplements (other than what is provided) and natural sources of astaxanthin including algae, yeast, salmon, trout, krill, shrimp and crayfish during the 10-week study.
* Categorized as "low risk" using the American College of Sports Medicine screening questionnaire.
* Generally healthy and without chronic disease including cardiovascular disease (e.g., heart disease, stroke), cancer, type 1 and 2 diabetes, rheumatoid arthritis.

Exclusion Criteria:

* Inability to comply with study requirements.
* Body weight below 110 pounds.
* Pregnant or breastfeeding.
* Any other concurrent condition which, in the opinion of the primary investigator (PI), would preclude participation in this study or interfere with compliance.
* Current diagnosis of cardiovascular disease, diabetes, or cancer (except for non-melanoma skin cancer).
* History of allergic reactions to astaxanthin.
* Using drugs with 5-alpha-reductase inhibitor (Proscar, Propecia, Avodart, Jalyn).

Ages: 18 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Plasma lipid mediators | Change from pre-study to post-4 weeks supplementation, and immediately post-exercise, and 1.5 hours-, 3 hours-, and 24 hours-post-exerciseingestion to 8- and 24-hours post-ingestion
  Plasma concentrations of arachadonic acid oxidized derivatives from LC-MS-MS analysis

SECONDARY OUTCOMES:
Plasma proteins | Change from pre-study to post-4 weeks supplementation, and immediately post-exercise, and 1.5 hours-, 3 hours-, and 24 hours-post-exerciseingestion to 8- and 24-hours post-ingestion
  Plasma concentrations of immune- and inflammation-related proteins from proteomics profiling using LC-MS-MS analysis
Plasma cytokine panel | Change from pre-study to post-4 weeks supplementation, and immediately post-exercise, and 1.5 hours-, 3 hours-, and 24 hours-post-exerciseingestion to 8- and 24-hours post-ingestion
  Plasma concentrations of cytokines most influenced by exercise inclduing IL6, IL8, IL10, MCP-1, IL1ra, GCSF

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share data upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: September 2022; indefinitely
Access Criteria: Upon request